CLINICAL TRIAL: NCT04860427
Title: Trapezoidal Condylar Plate (TCP) Versus Two Miniplates in Treatment of Subcondylar Fracture
Brief Title: Trapezoidal Condylar Plate (TCP) in Treatment of Subcondylar Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, mona oraby, Assistant lecturer, oral and maxillofacial surgery department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB NO 00010556-IORG 0008839
Record Dates: First submitted 2021-04-08; First posted 2021-04-27 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Fracture of Condylar Process

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trapezoidal condylar plate (Active Comparator): Trapezoidal condylar plate open reduction and internal fixation of subcondylar fractures
  Interventions: Device: trapezoidal condylar plate
- two miniplates (Active Comparator): two miniplates open reduction and internal fixation of subcondylar fractures
  Interventions: Device: two miniplates

INTERVENTIONS:
Device: trapezoidal condylar plate — trapezoidal condylar plate open reduction and fixation
  Arms: Trapezoidal condylar plate
Device: two miniplates — two miniplates open reduction and fixation
  Arms: two miniplates

SUMMARY:
Background: Condylar fracture is a common mandibular fracture which accounts for 25-40%. Nowadays the preference started to change towards open reduction because of the late complications that might happen in case of closed treatment.

A Transmasseteric Anteroparotid (TMAP) approach for open reduction and internal fixation of condylar fractures overcomes the problems of difficult access and facial nerve injury risk of other conventional approaches.

Different plating options are available for internal fixation of the condyle and subcondylar region. Trapezoidal Condylar Plates (TCP) specifically developed for the osteosynthesis of low and high subcondylar fracture. These plates were designed to closely follow the tensile strain lines along the rim of the sigmoid notch anteriorly combined with a posterior arm to parallel the condylar axis free of harmful bending strains.

DETAILED DESCRIPTION:
Background: Condylar fracture is a common mandibular fracture which accounts for 25-40%. It is the most controversial fractures regarding diagnosis and management.

For several years, closed reduction has been preferred over open reduction to avoid surgical complications. Nowadays the preference started to change towards open reduction because of the late complications that might happen in case of closed treatment.

A Transmasseteric Anteroparotid (TMAP) approach for open reduction and internal fixation of condylar fractures overcomes the problems of difficult access and facial nerve injury risk of other conventional approaches.

Different plating options are available for internal fixation of the condyle and subcondylar region. Trapezoidal Condylar Plates (TCP) specifically developed for the osteosynthesis of low and high subcondylar fracture. These plates were designed to closely follow the tensile strain lines along the rim of the sigmoid notch anteriorly combined with a posterior arm to parallel the condylar axis free of harmful bending strains.

Aim: Our aim in this study is to assess the use of TCP in the subcondylar fracture in comparison to the use of conventional two miniplates method.

Materials and methods: This prospective randomized clinical trial will enroll 20 patients with subcondylar fracture indicated for open reduction and internal fixation. Group A will undergo fixation with TCP and group B will have two miniplates fixation. Both groups will have Transmasseteric Anteroparotid approach.

Results: The results of the two groups will be compared clinically and radiographically.

Keywords: Subcondylar fracture, Trapezoidal condylar plate, two miniplates, open treatment for condyle, geometric subcondylar plates, transmasseteric anteroparotid approach.

ELIGIBILITY:
Inclusion Criteria:

* 1- Medically fit patients free from relevant conditions that contraindicate surgery.

  2- Patients with age ranged from 20-40 years old. 3- Patients suffering from displaced extracapsular mandibular subcondylar fracture indicated for open reduction including Difficulty of obtaining adequate occlusion by closed method, Radiological signs of the following
  1. Deviation of the fragment from the axis of the ascending ramus in medial or lateral direction more than 10°.(22)
  2. Shortening of the ascending ramus ≥ 2 mm measured from the roof of glenoid fossa to the inferior border of the ascending ramus of the mandible.(22)
  3. Dislocation of the condyle from the glenoid fossa.(48)

     Exclusion Criteria:
* 1. Patients who were not able to follow the information given or to make a decision themselves due to mental or other problems.

  2. Any absolute contraindication for surgery. 3. Patient with undisplaced condylar fractures that doesn't cause malocclusion or loss of facial heightening and can be treated conservatively.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
comparison of functional mandibular movement between the two groups | preopertive, 1 week, 1month , 3 months , 6months
  the change mandibular movement in mm
comparison of occlusion between the two groups | preopertive, 1 week, 1month , 3 months , 6months
  the change in occlusion intercuspation assessed visually by the surgeon and by asking the patient
comparison of helikmo index between the two groups | preopertive, 1 week, 1month , 3 months , 6months
  the change in helikmo index score
comparison in pain between the two groups | preopertive, 1 week, 1month
  the change in pain value with Visual analogue Scale With a visual analogue scale (VAS) with values from 0 (no pain) to 10 (strongest pain or discomfort)
comparison in ramus height shortening between the two groups | 1 day, 3 months, 6 months.
  radiographically: assess the adequacy of reduction by th change in ramus height in mm
comparison in condylar angulation between the two groups | 1 day, 3 months, 6 months.
  radiographically: assess the adequacy of reduction by measuring the change in condylar angulation
bone density change comparison between the two groups | 1 day postoperative, 1month and 3months
  assessment with CT in Hounsfield value measurements.

SECONDARY OUTCOMES:
Transmasseteric Anteroparotid surgical approach | intraopertive
  To evaluate the Transmasseteric Anteroparotid surgical approach for the subcondylar fracture regarding the time taken to reach the fracture line and convenience of the approach.
the stress on plates by using finite element analysis | immediate postopertive
  stress values (Mpa) were obtained in this study for each of the two models during load application
the displacement (micromotion) | immediate postoperative
  the amount of vertical displacement induced around the fracture surface (µm)

CONTACTS AND LOCATIONS:
Overall Officials: nagy el prince, professor, Study Chair — oral and maxillofacial surgery, alexanderia university
Locations (1):
- Mona Oraby, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No